CLINICAL TRIAL: NCT04174222
Title: The Effect of Deep Neuromuscular Blockade During Robotic Assisted Radical Prostatectomy on Intraoperative Respiratory Mechanics and Postoperative Pulmonary Complications : a Prospective Randomized Controlled Trial
Brief Title: The Effect of Deep Neuromuscular Blockade on Respiratory Mechanics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chang-Hoon Koo, Assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RALP-PIP
Record Dates: First submitted 2019-11-21; First posted 2019-11-22 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Neuromuscular Blockade

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate block (Active Comparator): 5-10mg rocuronium is administered to maintain train-of-four count 1-2. At the end of surgery, sugammadex 2mg/kg is administered IV for reversal of neuromuscular block.
  Interventions: Other: Moderate NMB
- Deep block (Experimental): 5-10mg rocuronium is administered to maintain train-of-four count 0, and post tetanic count 1-2 (deep block). At the end of surgery, sugammadex 4 mg/kg are administered IV for reversal of neuromuscular block
  Interventions: Other: Deep NMB

INTERVENTIONS:
Other: Moderate NMB — Neuromuscular block was maintained at train of four count 1-2.
  Arms: Moderate block
Other: Deep NMB — Neuromuscular block was maintained at train of four count 0 and post-tetanic count1-2.
  Arms: Deep block

SUMMARY:
This study is a randomized, controlled, double-blinded, and parallel design study. A total 58 patients were randomized to receive a deep block or a moderate block scheduled for elective robot assisted laparoscopic radical prostatectomy. Intraoperative peak inspiratory pressure and plateau pressure are assessed.

DETAILED DESCRIPTION:
Patients >18 years of age with an america society of anesthesiologist classification of I or II who are scheduled to undergo elective robot assisted laparoscopic radical prostatectomy are included. The exclusion criteria are a history of neuromuscular, renal, or hepatic disease, known allergy to rocuronium or sugammadex. Patients are randomized to either the moderate or deep neuromuscular blockade group using Random Allocation Software (version 1.0). In the operating room, routine monitoring is performed, including electrocardiography, non-invasive arterial pressure measurements, and pulse oximetry. Additionally, acceleromyography are applied to monitor the response of the adductor pollicis muscle. After the induction of anesthesia with propofol and before rocuronium administration, the TOF-Watch-SX is calibrated and stabilised, and a series of train-of-four (TOF) measurements are documented every 1 min. Next, intravenous rocuronium at 0.6 mg/kg was administered, and tracheal intubation was performed after confirmation of relaxation. Anesthesia is maintained with desflurane and target-controlled infusion of remifentanil while monitoring the bispectral index. Intravenous rocuronium (5-10 mg) is used to maintain moderate (TOF count of 1 or 2) or deep (post-tetanic count [PTC] of 1 or 2) neuromuscular blockade. Peak inspiratory pressure and plateau pressure are recorded until 1 hour after pneumoperitoneum. At the end of the operation, the surgeon rated the surgical condition on a 5-point scale. Patients are reversed with intravenous sugammadex at 2 or 4 mg/kg. Postoperative pulmonary complications (SpO2 <100%, RR<8, atelectasis) are assessed and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo elective robot assisted radical prostatectomy,
* American Society of Anesthesiologists grade 1 or 2

Exclusion Criteria:

* Refuse to participate to the study
* history of neuromuscular diseases
* known allergy to rocuronium, sugammadex
* patients scheduled for intensive care unit transfer
* Body Mass Index > 30 kg/m2
* Severe renal function impairment
* Moderete or severe obstructive/restrictive lung disease

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Peak inspiratory pressure | until 1 hour after pneumoperitoneum
  measured through ventilator

SECONDARY OUTCOMES:
plateau pressure | until 1 hour after pneumoperitoneum
  measured through ventilator
dynamic lung compliance | until 1 hour after pneumoperitoneum
  Tidal volume/(Peak inspiratory pressure - PEEP)
static lung compliance | until 1 hour after pneumoperitoneum
  Tidal volume/(Plateau pressure - PEEP)
5-point surgical rating scale | 1 min at the end of surgery
  Rated by the surgeon who is in charge of the patient's operation and is blind to the patient's group assignment. (1 = excellent, 2 = good, 3 = acceptable, 4 = poor, 5 = extremely poor)
Postoperative pulmonary complications | postoperative 30 min
  SpO2 <90% or RR < 8/min, atelectasis confirmed by Chest X ray

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Hoon Koo, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No